CLINICAL TRIAL: NCT01518465
Title: A Phase 2 Study of Lenalidomide and Low-dose Dexamethasone in Combination With Dalteparin in Previously Untreated Multiple Myeloma
Brief Title: Dalteparin, Lenalidomide, and Low-Dose Dexamethasone in Treating Patients With Previously Untreated Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16M-11-1; NCI-2011-03784 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dalteparin; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (5000 IU dalteparin) (Experimental): Patients receive a prophylactic dose of dalteparin SC on days 1-28; lenalidomide PO on days 1-21; and low-dose dexamethasone PO on days 1, 8, 15, and 22.
  Interventions: Drug: dalteparin; Drug: lenalidomide; Drug: dexamethasone; Other: laboratory biomarker analysis
- Arm II (200 IU/kg dalteparin) (Experimental): Patients receive a therapeutic dose of dalteparin SC on days 1-21 and lenalidomide PO and low-dose dexamethasone PO as in Arm I.
  Interventions: Drug: dalteparin; Drug: lenalidomide; Drug: dexamethasone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dalteparin — Given SC
  Other Names: DAL; dalteparin sodium; Fragmin
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot phase II trial studies how well giving dalteparin, lenalidomide, and low-dose dexamethasone together works in treating patients with previously untreated multiple myeloma. Anticoagulants, such as dalteparin, may help prevent blood clots from forming in patients being treated with lenalidomide and dexamethasone for multiple myeloma. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving dalteparin, lenalidomide, and dexamethasone together may be an effective treatment for multiple myeloma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To select a dose of Dalteparin to be used with Lenalidomide and low-dose dexamethasone in future trials for patients with previously untreated multiple myeloma (MM), based on toxicity, selected biomarkers (M-spike, interleukin [IL]-6) related to response and other markers of coagulation.

SECONDARY OBJECTIVES:

I. To evaluate overall response rate (ORR = complete response [CR] + partial response [PR]), and time to progression (TTP) for this regimen at each of the two Dalteparin doses.

II. To evaluate the safety profile of this regimen in untreated MM patients, at each of the two Dalteparin doses.

III. To study the effect of Dalteparin alone, and in combination with lenalidomide/dexamethasone on serum biomarkers of multiple myeloma (MM) and thrombosis.

IV. To explore possible associations between the ORR and incidence of venous thromboembolism (VTE) with serial syndecan-1, IL-6, tyrosine aminotransferase (TAT), D-dimer, P-selectin levels.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive a prophylactic dose of dalteparin subcutaneously (SC) on days 1-28; lenalidomide orally (PO) on days 1-21; and low-dose dexamethasone PO on days 1, 8, 15, and 22.

ARM II: Patients receive a therapeutic dose of dalteparin SC on days 1-21 and lenalidomide PO and low-dose dexamethasone PO as in Arm I.

In both arms, treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with residual responding disease may receive 2 additional courses. After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of active MM requiring treatment, as diagnosed by a bone marrow biopsy within 8 weeks prior to study enrollment
* Patients must not have received any previous treatment for MM (localized radiation therapy or single agent pulse steroid therapy for acute MM crises is permitted)
* Life expectancy of greater than 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky >= 50%)
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Transaminases (aspartate aminotransferase [AST]/alanine aminotransferase [ALT]) < 2.5 x ULN
* Alkaline phosphatase < 2.5 ULN
* Platelets >= 75,000 cells/mm3
* Hemoglobin >= 8.0 g/dL
* Absolute neutrophil count (ANC) > 1,000 cells/mm3 NOTE: Patients with platelet count < 75,000 or hemoglobin < 8.0 g/dl,or ANC <1,000 cell/mm3 secondary to extensive bone marrow disease can be enrolled at Principal Investigator's (PI) discretion with appropriate transfusion and/or cytokine support
* Creatinine =< 2.5 mg/dL (=< 200 mmol/L) or creatinine clearance > 30 ml/min (as calculated by the Cockcroft-Gault formula)
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10-14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* Willingness and ability to sign informed consent for the clinical trial

Exclusion Criteria:

* Patients who have had any prior chemotherapy for MM; with the exception of pulse steroids for any myeloma-related acute events
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational
* Pregnant or lactating women
* Active serious infections uncontrolled by antibiotics at the time of treatment initiation
* Inability to give voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Failure to comply with birth control methods as described above
* Any serious medical or psychiatric condition or reason that, in the PI's opinion, makes the patient unsuitable to participate in this clinical trial
* Known to be human immunodeficiency virus (HIV) positive (if the status of HIV is not known and patient is not at risk, as determined by the PI, then the patient will not be specifically tested for HIV); HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with lenalidomide and/or dalteparin. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer (organ-confined, early stage disease) after curative therapy
* Patients with M protein >6 gm/dl prior to starting treatment will be excluded from the initial "run-in" cohort on both arms of the study, but will be eligible for the subsequent enrollment of patients who do not have a run-in phase with dalteparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who experienced grade 4 hemorrhage regardless of attribution, or grade 3 hemorrhage that is possibly, probably, or definitely attributable to dalteparin (Arm II) | Up to 2 years

SECONDARY OUTCOMES:
Toxicities observed at each dose level, in terms of type (organ affected, laboratory determination), severity (by Common Toxicity Criteria [CTC]) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mohrbacher, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States